CLINICAL TRIAL: NCT01663831
Title: Repellents as Added Control Measure to Long Lasting Insecticidal Nets to Target the Residual Transmission in Southeast Asia: a Step Forwards to Malaria Elimination
Brief Title: Repellents as Added Control Measure to Long Lasting Insecticidal Nets
Acronym: MalaResT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Institute of Tropical Medicine, Belgium (Other)
Collaborators: NCHADS - Ministry of Health of Cambodia (Other); Institut Pasteur (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: OPP1032354
Record Dates: First submitted 2012-07-17; First posted 2012-08-13 (Estimated); Last update posted 2025-05-11 (Actual); Status verified 2025-05

CONDITIONS: Malaria
Keywords: Outdoor Malaria Transmission; Anopheles; Topical repellent; Early biting vector; Long Lasting Insecticidal Net (LLIN); Cambodia
MeSH Terms: conditions — Malaria

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Topical Repellent & LLIN (Experimental)
  Interventions: Other: Mosquito topical repellent
- Long Lasting Insecticidal Nets (No Intervention): Brand Name LLIN: Olyset Net
  Active ingredient: permethrin

INTERVENTIONS:
Other: Mosquito topical repellent — Daily repellent use, before and after sleeping hours during the malaria season (6 months) in addition to the use of Long Lasting Insecticidal Nets during sleeping hours.
  Other Names: Brand name: Autan; Active ingredient: Icaridin
  Arms: Topical Repellent & LLIN

SUMMARY:
The scaling up of Long Lasting Insecticidal Nets (LLIN) and the expansion of Indoor Residual Spraying (IRS) has contributed to a significant decrease of malaria worldwide. However these control methods tackle only indoor and night biting vectors. The proportion of transmission occurring outdoors and before sleeping hours or so-called "residual transmission" is steadily increasing and may compromise the effort towards malaria elimination.

The purpose of this study is to raise evidence on the effectiveness of mass use of topical repellents in addition to LLINs in controlling malaria infections.

A multidisciplinary approach will be used to collect information on the most important factors that contribute to the successful reduction of "residual malaria transmission". In a first objective the epidemiological efficacy of repellents on prevalence of malaria carriers and malaria incidence will be assessed. To achieve this goal 98 communities will be randomly assigned to one of two treatment arms (LLIN and LLIN + repellent). Within a community a cross sectional random sample of 65 people will be drawn at the beginning and the end of the malaria season to obtain an estimate of the malaria prevalence. The second objective will handle the entomological efficacy and persistence of the topical repellent on malaria vectors. And lastly the acceptability, adherence and adequacy of the topical repellents will be studied in a third objective.

ELIGIBILITY:
Inclusion Criteria:

* All household members volunteering from selected communities

Exclusion Criteria:

* Infants less than 2 years

Min Age: 2 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 40000 (Actual)
Dates: Start 2012-05; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Change from baseline in malaria prevalence at 6 months | 6 months
  Malaria prevalence (PCR detection) will be measured in both study arms at the start and end of the malaria season for 2 consecutive years.

SECONDARY OUTCOMES:
Malaria incidence | 6 months
  Through passive RDT case detection

CONTACTS AND LOCATIONS:
Overall Officials: Marc Coosemans, Professor, Principal Investigator — Institute of Tropical Medicine Antwerp
Locations (1):
- Banlung, Ratanakiri, Cambodia

REFERENCES:
- [Derived] Sluydts V, Durnez L, Heng S, Gryseels C, Canier L, Kim S, Van Roey K, Kerkhof K, Khim N, Mao S, Uk S, Sovannaroth S, Grietens KP, Sochantha T, Menard D, Coosemans M. Efficacy of topical mosquito repellent (picaridin) plus long-lasting insecticidal nets versus long-lasting insecticidal nets alone for control of malaria: a cluster randomised controlled trial. Lancet Infect Dis. 2016 Oct;16(10):1169-1177. doi: 10.1016/S1473-3099(16)30148-7. Epub 2016 Jun 29. PMID 27371977
- [Derived] Heng S, Durnez L, Gryseels C, Van Roey K, Mean V, Uk S, Siv S, Grietens KP, Sochantha T, Coosemans M, Sluydts V. Assuring access to topical mosquito repellents within an intensive distribution scheme: a case study in a remote province of Cambodia. Malar J. 2015 Nov 24;14:468. doi: 10.1186/s12936-015-0960-4. PMID 26597653
- [Derived] Canier L, Khim N, Kim S, Sluydts V, Heng S, Dourng D, Eam R, Chy S, Khean C, Loch K, Ken M, Lim H, Siv S, Tho S, Masse-Navette P, Gryseels C, Uk S, Van Roey K, Grietens KP, Sokny M, Thavrin B, Chuor CM, Deubel V, Durnez L, Coosemans M, Menard D. An innovative tool for moving malaria PCR detection of parasite reservoir into the field. Malar J. 2013 Nov 9;12:405. doi: 10.1186/1475-2875-12-405. PMID 24206649